CLINICAL TRIAL: NCT05216315
Title: Non-invasive Transcranial Direct Current Stimulation to Improve Cognitive Efficiency
Brief Title: tDCS and Cognitive Efficiency in Ageing
Acronym: FRtDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Juan Carlos Melendez, Coordinator of Doctoral Programme in Psychogerontology: Life Cycle Perspective, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1526539449220
Record Dates: First submitted 2022-01-19; First posted 2022-01-31 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Aging; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: sham versus stimulation
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS. Transcranial direct current stimulation (Experimental): The stimulation time was 20 minutes, with an initial and final ramp of 30 seconds so that the participant could adapt to the sensation of the current. 10 sessions. Constant current intensity of 2 mA The anode was placed on position F3, coinciding with the dorsolateral prefrontal cortex, and the cathode was placed on Fp2, coinciding with the right supraorbital area (rSO).
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham stimulation (Sham Comparator): The sham group received direct current only on the ramps to generate a sensation of the effect.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — 10 sessions of tDCS stimulation on dorsolateral prefrontal cortex with the apparatus HDC stimulator (Newronika TM)
  Other Names: Transcranial direct current stimulation
  Arms: tDCS. Transcranial direct current stimulation
Device: Sham stimulation — The sham group received direct current only on the ramps to generate a sensation of the effect.10 sessions
  Other Names: Transcranial direct current stimulation
  Arms: Sham stimulation

SUMMARY:
Normal aging is associated with a progressive decline in cognitive functions, especially memory. This decline in cognitive function can negatively impact the quality of life of older adults. Although there are currently few possibilities to prevent and/or slow the signs of cognitive decline, both those associated with age and neurodegenerative pathologies, one of the non-invasive brain stimulation techniques that has gained attention in recent years is Transcranial Direct Current Stimulation (tDCS). tDCS is a technique based on the application of a low-intensity (< 2 mA) direct electrical current between two large-area electrodes placed on various surface areas of the head. Moreover, according to safety-related meta-analyses it is a very safe technique, without any major side effects, provided that internationally established safety protocols are taken into account in its application. This technique has recently been investigated as a potential treatment for both healthy elderly people and people with mild cognitive impairment and Alzheimer's disease in several cognitive variables, having shown encouraging results in working memory learning curves, modulation of plasticity and recognition tasks. This project aims to implement an intervention using transcranial direct current stimulation in healthy older adults, MCI and AD. The main objective is to test if there is an improvement in cognitive efficiency and if the changes are maintained over time (1 month). For this purpose, the effect of the technique will be studied on participants assigned to treatment and control groups, analyzing the possible modifications in the following cognitive variables: cognitive plasticity and learning potential, recognition and familiarity and false alarms.

DETAILED DESCRIPTION:
The clinical trial protocol involves the recruitment of participants from three different groups: healthy older adults, individuals with mild cognitive impairment (MCI), and patients with Alzheimer's disease (AD). Participants will be randomly assigned to either a treatment group or a control group.

For the treatment group, transcranial direct current stimulation (tDCS) will be administered over a specified period using a standard protocol involving the application of low-intensity electrical current (< 2 mA) through electrodes placed on specific scalp areas. The duration and frequency of stimulation will be predetermined based on scientific literature and established safety recommendations.

The control group will receive a sham procedure where a low-intensity current, having no effect on neuronal activity, will be applied to maintain treatment masking.

Prior to commencing the intervention, a baseline assessment of participants' cognitive functions will be conducted using a battery of standardized tests, including measures of cognitive plasticity, memory, attention, executive functions, and other relevant cognitive abilities.

During the intervention period, regular tDCS or placebo sessions will be conducted according to participants' assigned groups. Additionally, data on potential side effects and tolerability of the technique will be collected.

At the end of the intervention period, a post-treatment assessment will be conducted to determine any changes in participants' cognitive functions. These data will be compared to baseline assessments to ascertain the intervention's efficacy.

Furthermore, participants will be followed up for a period of at least one month after the intervention to evaluate the persistence of effects and any potential long-term effects.

It is important to emphasize that this protocol will adhere to all ethical and safety regulations established by relevant regulatory authorities and ethics committees. Participants will be fully informed about the procedures and risks involved, and their informed consent will be obtained before their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

For the group of healthy older adults:

* MEC score greater than 26 points.
* GDS between 1 and 3.

For the MCI group:

* MEC score between 21 and 26 points.
* GDS between 1 and 3.

For the mild EA group:

* MEC score between 18 and 23 points.
* GDS between 3 and 4.

Exclusion Criteria:

* Presentation of contraindications to tDCS (presence of intracranial metal implants, intracranial hypertension, comitial risk).
* Significant asymptomatic neurovascular disease
* History of previous symptomatic stroke
* Alcohol or drug abuse/dependence
* Severe psychiatric symptoms
* Depressive symptoms higher than mild

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan C Melendez, Principal Investigator — University of Valencia
Locations (1):
- Faculty of Psychology, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
All the information of the study, as well as its results, will be shared in scientific publications and conferences related to the research area.
  The information that is intended to be published in scientific journals includes:
  1) Study Protocol, 2) Statistical Analysis, 3) Informed Consent Form, 4) Clinical Study Results.

REFERENCES:
- [Background] Dedoncker J, Brunoni AR, Baeken C, Vanderhasselt MA. A Systematic Review and Meta-Analysis of the Effects of Transcranial Direct Current Stimulation (tDCS) Over the Dorsolateral Prefrontal Cortex in Healthy and Neuropsychiatric Samples: Influence of Stimulation Parameters. Brain Stimul. 2016 Jul-Aug;9(4):501-17. doi: 10.1016/j.brs.2016.04.006. Epub 2016 Apr 12. PMID 27160468
- [Background] Deldar Z, Rustamov N, Blanchette I, Piche M. Improving working memory and pain inhibition in older persons using transcranial direct current stimulation. Neurosci Res. 2019 Nov;148:19-27. doi: 10.1016/j.neures.2018.12.007. Epub 2019 Jan 4. PMID 30615905
- [Background] Galli G, Vadillo MA, Sirota M, Feurra M, Medvedeva A. A systematic review and meta-analysis of the effects of transcranial direct current stimulation (tDCS) on episodic memory. Brain Stimul. 2019 Mar-Apr;12(2):231-241. doi: 10.1016/j.brs.2018.11.008. Epub 2018 Nov 17. PMID 30503376
- [Background] Hill AT, Fitzgerald PB, Hoy KE. Effects of Anodal Transcranial Direct Current Stimulation on Working Memory: A Systematic Review and Meta-Analysis of Findings From Healthy and Neuropsychiatric Populations. Brain Stimul. 2016 Mar-Apr;9(2):197-208. doi: 10.1016/j.brs.2015.10.006. Epub 2015 Oct 23. PMID 26597929
- [Background] Huo L, Zheng Z, Huang J, Li R, Li J, Li J. Transcranial Direct Current Stimulation Enhances Episodic Memory in Healthy Older Adults by Modulating Retrieval-Specific Activation. Neural Plast. 2020 Dec 5;2020:8883046. doi: 10.1155/2020/8883046. eCollection 2020. PMID 33354206
- [Background] Nissim NR, O'Shea A, Indahlastari A, Kraft JN, von Mering O, Aksu S, Porges E, Cohen R, Woods AJ. Effects of Transcranial Direct Current Stimulation Paired With Cognitive Training on Functional Connectivity of the Working Memory Network in Older Adults. Front Aging Neurosci. 2019 Dec 16;11:340. doi: 10.3389/fnagi.2019.00340. eCollection 2019. PMID 31998111
- [Background] Perceval G, Martin AK, Copland DA, Laine M, Meinzer M. Multisession transcranial direct current stimulation facilitates verbal learning and memory consolidation in young and older adults. Brain Lang. 2020 Jun;205:104788. doi: 10.1016/j.bandl.2020.104788. Epub 2020 Mar 19. PMID 32199339
- [Background] Summers JJ, Kang N, Cauraugh JH. Does transcranial direct current stimulation enhance cognitive and motor functions in the ageing brain? A systematic review and meta- analysis. Ageing Res Rev. 2016 Jan;25:42-54. doi: 10.1016/j.arr.2015.11.004. Epub 2015 Nov 30. PMID 26607412

RESULTS

PARTICIPANT FLOW:
Groups:
- tDCS. Transcranial Direct Current Stimulation: The stimulation time was 20 minutes, with an initial and final ramp of 30 seconds so that the participant could adapt to the sensation of the current. 10 sesions. Constant current intensity of 2 mA The anode was placed on position F3, coinciding with the dorsolateral prefrontal cortex, and the cathode was placed on Fp2, coinciding with the right supraorbital area (rSO).
  Transcranial direct current stimulation (tDCS): 10 sessions of tDCS stimulation on dorsolateral prefrontal cortex with the apparatus HDC stimulator (Newronika TM)
Period: Overall Study
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
Started | 19 | 19
Completed | 17 | 16
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (5.7) | 73.4 (6.2) | 75 (6.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 16 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Complutense Verbal Learning Test (TAVEC) - Memory
Description: This test presents a list of 16 words that, after being read by the evaluator, have to be repeated by the participant. The list is repeated five times (trials); the participant is again asked to remember the 16 words. The test was administered to evaluate the participant's immediate memory (Trial 1), learning ability (Trial 5 ). Post-intervention minus baseline. Scale is scored 0-16. Difference score range is (-16 to 16) with positive scores reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- tDCS. Transcranial Direct Current Stimulation: The stimulation time was 20 minutes, with an initial and final ramp of 30 seconds so that the participant could adapt to the sensation of the current. 10 sesions. Constant current intensity of 2 mA The anode was placed on position F7, coinciding with the dorsolateral prefrontal cortex, and the cathode was placed on Fp2, coinciding with the right supraorbital area (rSO).
  Transcranial direct current stimulation (tDCS): 10 sessions of tDCS stimulation on dorsolateral prefrontal cortex with the apparatus HDC stimulator (Newronika TM)
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 16
units on a scale
  Trial 1 | 0.94 (0.35) | -0.81 (0.03)
  Trial 5 | 1.65 (0.5) | -0.31 (0.4)

2. Primary Outcome: Digits Wechsler Intelligence Scale for Adults-III (WAIS-III)
Description: Direct and inverse digits of the Wechsler Intelligence Scale for Adults-III (Wechsler, 2001). These tests assess attentional capacity by exposing the participant to increasing amounts of information. On the direct digits task, which is used to assess immediate recall, the subject must repeat the sequence of numbers in the same order in which they are read by the examiner. On the inverse digit task, which assesses working memory and mental flexibility, the subject must say the digits backwards from the way they were presented by the examiner. Both tests are evaluated in the same way, assigning one point for each correct item, with a maximum score of 16 for both tests. Post-intervention minus baseline. Difference score range is (-16 to 16) with positive scores reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 16
units on a scale
  Direct Digits | 1.35 (0.62) | -0.18 (0.84)
  Inverse digits | 0.17 (1.15) | -0.43 (0.05)

3. Primary Outcome: Mini Mental State Examination
Description: This is a screening test for general cognitive status. This test is evaluated on a maximum of 30 points. Participants with scores equal to or below 23 would be considered cognitively deficient. Post-intervention minus baseline. Scale is scored 0-30. Difference score range is (-30 to 30) with positive scores reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 16
score on a scale | 2.18 (0.03) | -0.44 (1.28)

4. Secondary Outcome: Barcelona Test (BT) - Ability to Access and Recall Elements From the Lexical and Semantic Store
Description: Barcelona Test assesses the ability to access and recall lexical and semantic items by means of two subtests: a. Semantic fluency: recall the highest number of words from the category 'animals' in one minute; b. Phonological fluency: recall the highest number of words beginning with the letter 'p' in three minutes. Minimum and maximum range for Semantic fluency and Phonological fluency: 0 to n (no upper limit). Method of calculation: Scores for each subtest are reported separately. No combined scores or averages between subtests are calculated. Interpretation: Good categorical recall is considered good when evoking more than 16 animals in 1 minute and good verbal fluency when evoking more than 19 words beginning with 'p' in 3 minutes. This test assesses the ability to access and recall items from the lexical and semantic store. Processes involved: processing speed, cognitive flexibility and working memory. Post-intervention less baseline with positive scores reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: Number of words evoked
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 16
Number of words evoked
  Semantic fluency | 0.47 (4.47) | -5.72 (4.22)
  Phonological fluency | 1.77 (0.1) | 0.69 (0.46)

5. Other Pre Specified Outcome: Global Deterioration Scale (GDS)
Description: This test is evaluated on a maximum of 30 points. Participants with scores equal to or below 23 would be considered cognitively deficient.
Time Frame: Baseline to approximately 4 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Memory Alteration Test (M@T) - Cognitive Impairment
Description: This test offers a rapid and effective screening with excellent discriminative properties for amnestic Mild Cognitive Impairment (MCI-A) and early AD in the general primary care population. The test assesses a variety of abilities such as encoding, orientation, semantic memory and free recall. It consists of oral questions with only one possible answer, and the maximum achievable score is 50 points. The optimal cut-off point for distinguishing amnestic-like mild cognitive impairment from subjective memory complaints is 37 points. The optimal cut-off point for Alzheimer's disease is 31 points. Post-intervention minus baseline. Scale is scored 0-50. Difference score range is (-50 to 50) with positive scores reflecting improvement.
Time Frame: Baseline to approximately 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
Number analyzed (Participants) | 17 | 18
score on a scale | 6.06 (2.19) | -0.88 (1.7)

7. Other Pre Specified Outcome: Experimental Task - Recognition Familiarity and False Alarms
Description: This experimental task is composed by three lists of words with two conditions: half and entire.
  The half condition included two lists of 50 words each, formed entirely from the following letters of the Spanish alphabet: a, e, u, b, d, g, j, n, r, and z (list A) or i, o, c, f, h, l, m, p, s, t, v, and y (list B).
  List C (entire condition) contained 50 words formed from the entire alphabet, with the only criterion being that each word had to contain at least one letter from list A and at least one letter from list B.
  In the half condition, the recognition estimates for each participant were derived by subtracting the proportion of false alarms on words with the same letters, as in the study list, from the proportion of hits, whereas in the entire condition, the recognition estimates were derived by subtracting the proportion of false alarms on words with all the letters in the alphabet from the proportion of hits as a way to control the response bias of the participants.
Time Frame: Baseline to approximately 4 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | tDCS. Transcranial Direct Current Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT05216315/Prot_SAP_000.pdf